CLINICAL TRIAL: NCT05017727
Title: Does Closed-loop Automated Oxygen Control During Mechanical Ventilation Reduce Hypoxic Events? A Randomised Controlled Crossover Study in Ventilated Infants
Brief Title: Closed-loop Oxygen Control in Ventilated Infants Born at or Near Term
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 298164
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Pre-Term; Respiratory Disease
MeSH Terms: conditions — Premature Birth; Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Closed-loop automated oxygen control with Oxygenie Auto-O2 software (SLE6000) — The 'Oxygenie' is a closed loop automated oxygen control system that has been incorporated into a software module for the SLE6000 infant ventilators. This software control system allows targeting SpO2 values by controlling FiO2.

SUMMARY:
Ventilated neonates frequently require supplementary oxygen to allow for adequate oxygen delivery to the tissues and normal cell metabolism. Oxygen treatment should be monitored carefully as both excessive and inadequate dosing can have detrimental effects for the infants. Hypoxia (giving too little oxygen) increases mortality and later disability whereas hyperoxia (giving too much oxygen) increases the risk of complications such as retinopathy of prematurity and lung disease. Although very preterm and low birth weight infants represent the majority of ventilated neonates, more mature infants may also require mechanical ventilation at birth and provision of supplementary oxygen. Therefore, they may suffer from complications related to hypoxia or hyperoxia. Hence, their oxygen saturation levels and the amount of the inspired oxygen concentration provided should be continuously monitored.

Oxygen control is traditionally monitored and adjusted manually by the nurse looking after the infant. Closed-loop automated oxygen control (CLAC) is a more recent approach that involves the use of a computer software incorporated into the ventilator. The software uses an algorithm that automatically adjusts the amount of inspired oxygen to maintain oxygen saturation levels in a target range. Evidence suggests that CLAC increases the time spent in the desired oxygen target range, decreases the duration of hypoxia and hyperoxia and reduces the number of manual adjustments required by clinical staff. However previous studies have been limited to very small infants. With this study the investigators aim to evaluate the effectiveness of CLAC in ventilated infants born at 34 weeks gestation and beyond. The achievement of oxygen saturation targets and the number of manual adjustments required will be compared between periods of CLAC and manual control in a cohort of patients that has not been included in previous studies and could also benefit from the intervention. The investigators will also evaluate if CLAC reduces investigations performed to ventilated babies(blood gases, X-rays).

DETAILED DESCRIPTION:
This will be a randomised controlled crossover study. The investigators aim to recruit a minimum of 31 ventilated infants born at 34 weeks completed gestation and above and admitted to the Neonatal Intensive Care Unit at King's College Hospital over one year. Participants will undergo two monitoring periods each lasting 12 hours (8:00am-20:00pm): one with standard manually controlled oxygen and one with closed-loop automated oxygen control. Randomisation will be used to determine whether the first period will be manual or closed-loop automated oxygen control. The two monitoring periods will take place on two consecutive days to allow for clinical conditions to remain as stable as possible.

Infants with known congenital cyanotic heart disease will be excluded from the study as well as those undergoing surgery or any planned procedures during the monitoring period.

Informed written consent will be requested from the parents or legal guardians of the infants and the attending Neonatal Consultant will be requested to verbally assent to the study.

Randomisation of eligible infants whose parents consent to the study will be performed using an online randomisation generator to determine whether the first monitoring period will be manual adjustment or closed-loop automated oxygen control ("intervention" period).

Patients will be ventilated using SLE6000 ventilators. Ventilation settings will be manually adjusted by the clinical team as per unit's protocol. During the intervention period, in addition to standard care, infants will be also connected to the OxyGenie closed-loop oxygen saturation monitoring software (SLE). This software uses oxygen saturations from the SpO2 probe attached to the neonate, fed into an algorithm, to automatically adjust the percentage of inspired oxygen to maintain oxygen saturations within the target range. Manual adjustments including the percentage of FiO2 will be allowed at any point during the study including the period of automated oxygen control if deemed appropriate by the clinical team. Oxygen saturation levels and automatic adjustments to the inspired oxygen concentration will be captured by the ventilator software. Manual adjustments will be recorded during both monitoring periods. In addition to data collected from the ventilator, medical notes will be reviewed to determine any adverse events or clinical interventions to participants during the study. The number of blood gas samples taken and chest radiographs performed during each monitoring period will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 34 weeks completed gestation and above requiring mechanical ventilation and admitted to King's NICU
* Any gender, ethnicity or other comorbidities

Exclusion Criteria:

* Preterm infants less than 34 weeks gestation
* Infants with cyanotic congenital heart disease
* Infants undergoing planned procedures or surgery during the monitoring period
* Infants on high frequency oscillatory ventilation (HFOV)

Min Age: 34 Weeks | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This will be a randomised controlled crossover study. We aim to recruit a minimum of 31 ventilated infants born at 34 weeks completed gestation and above and admitted to the Neonatal Intensive Care Unit at our hospital over one year.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
The decrease in the percentage of time spent in extremes of hypoxia | Over 24 hours
  That will be assessed by evaluating the infant's respiratory status.

SECONDARY OUTCOMES:
The increase in the percentage of time spent within target oxygen saturation ranges (94-98%) | Over 24 hours
  This will be assessed by evaluating the infant's respiratory status.
The reduction in the number of manual adjustments required to the inspired oxygen concentration | Over 24 hours
  That will be assessed by reviewing the infant's medical records
The reduction in the number of blood gases and chest radiographs | Over 24 hours
  That will be assessed by reviewing the infant's medical records

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, Professor, Principal Investigator — King's College Hospital/ King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Consortium on Safe Labor; Hibbard JU, Wilkins I, Sun L, Gregory K, Haberman S, Hoffman M, Kominiarek MA, Reddy U, Bailit J, Branch DW, Burkman R, Gonzalez Quintero VH, Hatjis CG, Landy H, Ramirez M, VanVeldhuisen P, Troendle J, Zhang J. Respiratory morbidity in late preterm births. JAMA. 2010 Jul 28;304(4):419-25. doi: 10.1001/jama.2010.1015. PMID 20664042
- [Background] Colin AA, McEvoy C, Castile RG. Respiratory morbidity and lung function in preterm infants of 32 to 36 weeks' gestational age. Pediatrics. 2010 Jul;126(1):115-28. doi: 10.1542/peds.2009-1381. Epub 2010 Jun 7. PMID 20530073
- [Background] Pike KC, Lucas JS. Respiratory consequences of late preterm birth. Paediatr Respir Rev. 2015 Jun;16(3):182-8. doi: 10.1016/j.prrv.2014.12.001. Epub 2014 Dec 8. PMID 25554628
- [Background] Clark RH. The epidemiology of respiratory failure in neonates born at an estimated gestational age of 34 weeks or more. J Perinatol. 2005 Apr;25(4):251-7. doi: 10.1038/sj.jp.7211242. PMID 15605071
- [Background] Gouyon JB, Ribakovsky C, Ferdynus C, Quantin C, Sagot P, Gouyon B; Burgundy Perinatal Network. Severe respiratory disorders in term neonates. Paediatr Perinat Epidemiol. 2008 Jan;22(1):22-30. doi: 10.1111/j.1365-3016.2007.00875.x. PMID 18173781
- [Background] Ramadan G, Paul N, Morton M, Peacock JL, Greenough A. Outcome of ventilated infants born at term without major congenital abnormalities. Eur J Pediatr. 2012 Feb;171(2):331-6. doi: 10.1007/s00431-011-1549-8. Epub 2011 Aug 11. PMID 21833494
- [Background] Angus DC, Linde-Zwirble WT, Clermont G, Griffin MF, Clark RH. Epidemiology of neonatal respiratory failure in the United States: projections from California and New York. Am J Respir Crit Care Med. 2001 Oct 1;164(7):1154-60. doi: 10.1164/ajrccm.164.7.2012126. PMID 11673202
- [Background] Walsh BK, Smallwood CD. Pediatric Oxygen Therapy: A Review and Update. Respir Care. 2017 Jun;62(6):645-661. doi: 10.4187/respcare.05245. PMID 28546370
- [Background] Baba L, McGrath JM. Oxygen free radicals: effects in the newborn period. Adv Neonatal Care. 2008 Oct;8(5):256-64. doi: 10.1097/01.ANC.0000338015.25911.8a. PMID 18827514
- [Background] Askie LM, Henderson-Smart DJ, Irwig L, Simpson JM. Oxygen-saturation targets and outcomes in extremely preterm infants. N Engl J Med. 2003 Sep 4;349(10):959-67. doi: 10.1056/NEJMoa023080. PMID 12954744
- [Background] Supplemental Therapeutic Oxygen for Prethreshold Retinopathy Of Prematurity (STOP-ROP), a randomized, controlled trial. I: primary outcomes. Pediatrics. 2000 Feb;105(2):295-310. doi: 10.1542/peds.105.2.295. PMID 10654946
- [Background] BOOST-II Australia and United Kingdom Collaborative Groups; Tarnow-Mordi W, Stenson B, Kirby A, Juszczak E, Donoghoe M, Deshpande S, Morley C, King A, Doyle LW, Fleck BW, Davis PG, Halliday HL, Hague W, Cairns P, Darlow BA, Fielder AR, Gebski V, Marlow N, Simmer K, Tin W, Ghadge A, Williams C, Keech A, Wardle SP, Kecskes Z, Kluckow M, Gole G, Evans N, Malcolm G, Luig M, Wright I, Stack J, Tan K, Pritchard M, Gray PH, Morris S, Headley B, Dargaville P, Simes RJ, Brocklehurst P. Outcomes of Two Trials of Oxygen-Saturation Targets in Preterm Infants. N Engl J Med. 2016 Feb 25;374(8):749-60. doi: 10.1056/NEJMoa1514212. Epub 2016 Feb 10. PMID 26863265
- [Background] Saugstad OD, Aune D. In search of the optimal oxygen saturation for extremely low birth weight infants: a systematic review and meta-analysis. Neonatology. 2011;100(1):1-8. doi: 10.1159/000322001. Epub 2010 Dec 9. PMID 21150224
- [Background] Williams LZJ, McNamara D, Alsweiler JM. Intermittent Hypoxemia in Infants Born Late Preterm: A Prospective Cohort Observational Study. J Pediatr. 2019 Jan;204:89-95.e1. doi: 10.1016/j.jpeds.2018.08.048. Epub 2018 Oct 1. PMID 30287066
- [Background] Lakshminrusimha S, Konduri GG, Steinhorn RH. Considerations in the management of hypoxemic respiratory failure and persistent pulmonary hypertension in term and late preterm neonates. J Perinatol. 2016 Jun;36 Suppl 2:S12-9. doi: 10.1038/jp.2016.44. PMID 27225960
- [Background] Askie LM, Darlow BA, Finer N, Schmidt B, Stenson B, Tarnow-Mordi W, Davis PG, Carlo WA, Brocklehurst P, Davies LC, Das A, Rich W, Gantz MG, Roberts RS, Whyte RK, Costantini L, Poets C, Asztalos E, Battin M, Halliday HL, Marlow N, Tin W, King A, Juszczak E, Morley CJ, Doyle LW, Gebski V, Hunter KE, Simes RJ; Neonatal Oxygenation Prospective Meta-analysis (NeOProM) Collaboration. Association Between Oxygen Saturation Targeting and Death or Disability in Extremely Preterm Infants in the Neonatal Oxygenation Prospective Meta-analysis Collaboration. JAMA. 2018 Jun 5;319(21):2190-2201. doi: 10.1001/jama.2018.5725. PMID 29872859
- [Background] Hagadorn JI, Furey AM, Nghiem TH, Schmid CH, Phelps DL, Pillers DA, Cole CH; AVIOx Study Group. Achieved versus intended pulse oximeter saturation in infants born less than 28 weeks' gestation: the AVIOx study. Pediatrics. 2006 Oct;118(4):1574-82. doi: 10.1542/peds.2005-0413. PMID 17015549
- [Background] Sink DW, Hope SA, Hagadorn JI. Nurse:patient ratio and achievement of oxygen saturation goals in premature infants. Arch Dis Child Fetal Neonatal Ed. 2011 Mar;96(2):F93-8. doi: 10.1136/adc.2009.178616. Epub 2010 Oct 30. PMID 21037284
- [Background] Dargaville PA, Sadeghi Fathabadi O, Plottier GK, Lim K, Wheeler KI, Jayakar R, Gale TJ. Development and preclinical testing of an adaptive algorithm for automated control of inspired oxygen in the preterm infant. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F31-F36. doi: 10.1136/archdischild-2016-310650. Epub 2016 Sep 15. PMID 27634820
- [Background] Dani C. Automated control of inspired oxygen (FiO2 ) in preterm infants: Literature review. Pediatr Pulmonol. 2019 Mar;54(3):358-363. doi: 10.1002/ppul.24238. Epub 2019 Jan 10. PMID 30632296
- [Background] Sturrock S, Ambulkar H, Williams EE, Sweeney S, Bednarczuk NF, Dassios T, Greenough A. A randomised crossover trial of closed loop automated oxygen control in preterm, ventilated infants. Acta Paediatr. 2021 Mar;110(3):833-837. doi: 10.1111/apa.15585. Epub 2020 Oct 6. PMID 32969040
- [Background] Sturrock S, Williams E, Dassios T, Greenough A. Closed loop automated oxygen control in neonates-A review. Acta Paediatr. 2020 May;109(5):914-922. doi: 10.1111/apa.15089. Epub 2019 Nov 27. PMID 31715041
- [Background] Chowdhury O, Wedderburn CJ, Lee S, Hannam S, Greenough A. Respiratory support practices in infants born at term in the United Kingdom. Eur J Pediatr. 2012 Nov;171(11):1633-8. doi: 10.1007/s00431-012-1784-7. Epub 2012 Jul 22. PMID 22821075
- [Background] Bhat P, Chowdhury O, Shetty S, Hannam S, Rafferty GF, Peacock J, Greenough A. Volume-targeted versus pressure-limited ventilation in infants born at or near term. Eur J Pediatr. 2016 Jan;175(1):89-95. doi: 10.1007/s00431-015-2596-3. Epub 2015 Aug 4. PMID 26239663
- [Background] Chowdhury O, Greenough A. Neonatal ventilatory techniques - which are best for infants born at term? Arch Med Sci. 2011 Jun;7(3):381-7. doi: 10.5114/aoms.2011.23400. Epub 2011 Jul 11. PMID 22295020
- [Background] Chowdhury O, Rafferty GF, Lee S, Hannam S, Milner AD, Greenough A. Volume-targeted ventilation in infants born at or near term. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F264-6. doi: 10.1136/archdischild-2011-301041. Epub 2011 Dec 22. PMID 22194469
- [Background] Reynolds PR, Miller TL, Volakis LI, Holland N, Dungan GC, Roehr CC, Ives K. Randomised cross-over study of automated oxygen control for preterm infants receiving nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F366-F371. doi: 10.1136/archdischild-2018-315342. Epub 2018 Nov 21. PMID 30464005